CLINICAL TRIAL: NCT02101814
Title: Analysis of Neuroendocrine Regulation of Balance Energy and Inflammatory Factors in Obese Adults Submitted to Bariatric Surgery
Brief Title: Energy Balance and Inflammation in Obese Adults Bariatric Surgery Follow-up
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Bárbara Dal Molin Netto, Energy balance and inflammatory parameters after RYGB, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BNetto
Record Dates: First submitted 2014-03-26; First posted 2014-04-02 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Obesity; Morbid Obesity; Metabolic Syndrome; Inflammation; Energy Balance
MeSH Terms: conditions — Obesity; Obesity, Morbid; Metabolic Syndrome; Inflammation | interventions — Gastric Bypass; Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bariatric surgery (Other): Roux-en-Y gastric bypass procedure is being performed by surgery in all patients in this study.
  Interventions: Procedure: Roux-en-Y gastric bypass (bariatric surgery)

INTERVENTIONS:
Procedure: Roux-en-Y gastric bypass (bariatric surgery)

SUMMARY:
The prevalence of obesity is steadily growing in many parts of the world in order to reach epidemic proportions. Changes in signaling pathways state of hunger and satiety contribute to the increase in obesity and metabolic syndrome. Currently, the white adipose tissue, also is considered a secretory tissue by producing numerous adipokines involved in a chronic state of inflammation, which may interfere with the neuroendocrine regulation of energy balance that affect the weight loss process. The bariatric surgery is recommended as the most effective tool in the treatment and control of morbid obesity. The study population will consist of patients undergoing bariatric surgery of type Roux-en-Y gastric bypass. The study was performed in Clinical Hospital of the Federal University of Paraná (UFPR). This is a prospective cohort study with follow up of 6 and 24 months. The aim of this study is to assess the effects of weight loss after bariatric surgery associated anthropometric characteristic, metabolic changes (glucose, cholesterol profile,hepatic enzymes, Fibroblast growth factor- 21(FGF-21), blood pressure), the profile of adipokines pro/anti-inflammatory (adiponectin, interleukin-6 (IL-6),interleukin-10 (IL-10), C reactive protein (CRP), plasminogen activator inhibitor-1 (PAI-1), tumor necrosis factor alpha (TNF-α), intercellular adhesion molecule-1 (ICAM-1), resistin, frizzled-related protein 5 (SFrp5) and neuroendocrine regulation of energy balance (leptin, neuropeptide Y (NPY) , alpha-melanocyte stimulating hormone (α-MSH), melanin-concentrating hormone (MCH) and agouti-related peptide (AgRP), as well as the quality of life in obese adults.

ELIGIBILITY:
Inclusion Criteria:

* Age range 20-59 years
* BMI ≥ 40 kg/m2
* BMI ≥ 35 kg/m2 with comorbidity recognised by National Institutes of Health.

Exclusion Criteria:

* Patients in use of insulin
* Patients in use of Immunosuppressant
* Anti-inflammatory and/or immunosuppressant therapies
* Any malignancy
* Chronic kidney or liver disease
* Obesity caused by an endocrine disorder
* Patients with psychiatric disorders
* Smoker or alcohol dependence
* Patients with rheumatoid arthritis and/or autoimmune

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in anthropometric, metabolic, energy balance parameters and inflammatory profile at 6 months | 6 months

SECONDARY OUTCOMES:
Change from baseline in anthropometric, metabolic, energy balance parameters and inflammatory profile at 24 months | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ana R Dâmaso, PhD, Study Director — Federal University of São Paulo
Locations (1):
- Hospital de Clínicas/Federal University of Paraná, Curitiba, Paraná, Brazil

REFERENCES:
- See also: Related Info — http://asmbs.org/
- See also: Related Info — http://www.sbcb.org.br/